CLINICAL TRIAL: NCT05680545
Title: Volatile Anesthetic Pharmacokinetics During Extracorporeal Membrane
Brief Title: Volatile Anesthetic Pharmacokinetics During Extracorporeal Membrane Oxygenation
Acronym: Vol-ECMO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Diana Morales Castro, Junior Attending, MSICU Toronto General Hospital, Principal Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-6007; 2022-2746 (Other Grant/Funding Number: PSI Foundation)
Record Dates: First submitted 2022-12-16; First posted 2023-01-11 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Failure
Keywords: Extracorporeal membrane oxygenation; Volatile anesthetics; Sedation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, open-label, pharmacokinetic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sevoflurane vaporized in ECMO machines (Experimental): Patients' sedation will be managed with sevoflurane-based anesthesia directly vaporized into the ECMO machine.
  Interventions: Other: Sevoflurane vaporized in ECMO machines

INTERVENTIONS:
Other: Sevoflurane vaporized in ECMO machines — Sevoflurane will be directly vaporized into the ECMO machine through the sweep gas.

SUMMARY:
The goal of this study is to design a pilot trial evaluating the safety, feasibility, pharmacokinetic modeling, and physiological effects of a volatile anesthetic, sevoflurane, directly administered in extracorporeal membrane oxygenation machines.

DETAILED DESCRIPTION:
Venovenous extracorporeal membrane oxygenation (VV-ECMO) is a life-saving therapy for catastrophic respiratory failure, including severe COVID-19. Optimal drug dosing in critically ill patients is challenging due to concomitant organ dysfunction, and with the addition of ECMO, the level of complexity significantly increases.

ECMO PK interactions with intravenous (IV) sedatives are complex and therapeutic failures are often encountered, highlighting the need for alternative sedation strategies. To overcome these limitations, volatile anesthetics are a potential solution for sedation and analgesia. Nevertheless, their use has been limited during ECMO support due to the low respiratory volumes associated with the lung-protective strategies, and the concerns of bioavailability given the compromised native lung function. The overarching aim of this project is to evaluate a strategy to mitigate the influence of ECMO on sedatives pharmacokinetics, using volatile anesthetics directly vaporized into ECMO oxygenators.

The study will consist of two phases: the ex-vivo trial an the in-vivo trial. For the ex-vivo trial, two ECMO circuits primed with Ringer's lactate will be used to design the dosing recommendations for the feasibility trial. Vaporized sevoflurane will be delivered directly into the membrane oxygenator with the ECMO gas and evacuated through the wall suction. Sevoflurane concentrations will be monitored with an infrared multi-gas analyzer sensor at the ECMO gas outlet. The test will be performed with different sweep flows and sevoflurane concentrations. Sevoflurane concentrations will be measured in the fluid to design a dosing model to conduct the in-vivo trial.

The in-vivo trial will be a prospective, single-center, open-label, pilot feasibility/PK study of 10 patients receiving venovenous ECMO (VV ECMO) in the Medical-Surgical Intensive Care Unit (MSICU) at the Toronto General Hospital. Following informed consent, these patients will be enrolled and managed with sevoflurane-based anesthesia directly delivered into the ECMO machine. During their ECMO run, samples will be taken and sevoflurane concentrations analyzed with headspace gas chromatography and mass spectrometry. Sedation scales, surrogates of respiratory dynamics and effort, and biotrauma inflammatory cytokines levels will be obtained at the same time.

ELIGIBILITY:
Inclusion Criteria:

adult patients expected to be on VV ECMO support for a time frame of more than 24 hours and receiving a sevoflurane-based sedation protocol.

Exclusion Criteria:

* lack of informed consent for participation
* pregnancy
* serum bilirubin > 150 μmol/L
* ongoing massive blood transfusion requirement (> 50% blood volume transfused in the previous 8 hours)
* therapeutic plasma exchange and/or renal replacement therapy in the preceding 24 hours
* expected death or withdrawal of life support in the next 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sevoflurane plasma concentrations | 7 days
  Plasma concentrations of sevoflurane will be measured with gas chromatography and mass spectrometry

SECONDARY OUTCOMES:
Percentage of sevoflurane in ECMO exhausted gas | 7 days
  The volume/volume percentage of sevoflurane will be measured with an infrared multi-gas analyzer sensor at the sweep gas outlet
Respiratory dynamics and respiratory effort | 7 days
  Driving pressure, occlusion pressure, and P0.1 pressures will be measured with the patients mechanical ventilator daily
Plasma levels of ventilator-induced lung injury biomarkers | 7 days
  As a surrogate for ventilator-induced lung injury, plasma levels of interleukins 6 and 8, and necrosis tumor factor will be measured daily
Required doses of sedative adjuvants | 7 days
  The doses of other sedatives and analgesics, including opioids, antipsychotics, benzodiazepines, ketamine and propofol will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Diana Morales Castro, MD, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McMullan V, Alston RP, Tyrrell J. Volatile anaesthesia during cardiopulmonary bypass. Perfusion. 2015 Jan;30(1):6-16. doi: 10.1177/0267659114531314. Epub 2014 Apr 14. PMID 24732827
- [Background] LaGrew JE, Olsen KR, Frantz A. Volatile anaesthetic for treatment of respiratory failure from status asthmaticus requiring extracorporeal membrane oxygenation. BMJ Case Rep. 2020 Jan 15;13(1):e231507. doi: 10.1136/bcr-2019-231507. PMID 31948977
- [Background] Fan E, Gattinoni L, Combes A, Schmidt M, Peek G, Brodie D, Muller T, Morelli A, Ranieri VM, Pesenti A, Brochard L, Hodgson C, Van Kiersbilck C, Roch A, Quintel M, Papazian L. Venovenous extracorporeal membrane oxygenation for acute respiratory failure : A clinical review from an international group of experts. Intensive Care Med. 2016 May;42(5):712-724. doi: 10.1007/s00134-016-4314-7. Epub 2016 Mar 23. PMID 27007108
- [Background] Cheng V, Abdul-Aziz MH, Roberts JA, Shekar K. Overcoming barriers to optimal drug dosing during ECMO in critically ill adult patients. Expert Opin Drug Metab Toxicol. 2019 Feb;15(2):103-112. doi: 10.1080/17425255.2019.1563596. Epub 2019 Jan 3. PMID 30582435
- [Background] Shekar K, Roberts JA, Mcdonald CI, Fisquet S, Barnett AG, Mullany DV, Ghassabian S, Wallis SC, Fung YL, Smith MT, Fraser JF. Sequestration of drugs in the circuit may lead to therapeutic failure during extracorporeal membrane oxygenation. Crit Care. 2012 Oct 15;16(5):R194. doi: 10.1186/cc11679. PMID 23068416
- [Background] Shekar K, Roberts JA, Mullany DV, Corley A, Fisquet S, Bull TN, Barnett AG, Fraser JF. Increased sedation requirements in patients receiving extracorporeal membrane oxygenation for respiratory and cardiorespiratory failure. Anaesth Intensive Care. 2012 Jul;40(4):648-55. doi: 10.1177/0310057X1204000411. PMID 22813493
- [Background] Bellgardt M, Ozcelik D, Breuer-Kaiser AFC, Steinfort C, Breuer TGK, Weber TP, Herzog-Niescery J. Extracorporeal membrane oxygenation and inhaled sedation in coronavirus disease 2019-related acute respiratory distress syndrome. World J Crit Care Med. 2021 Nov 9;10(6):323-333. doi: 10.5492/wjccm.v10.i6.323. eCollection 2021 Nov 9. PMID 34888158
- [Background] Rand A, Zahn PK, Schildhauer TA, Waydhas C, Hamsen U. Inhalative sedation with small tidal volumes under venovenous ECMO. J Artif Organs. 2018 Jun;21(2):201-205. doi: 10.1007/s10047-018-1030-9. Epub 2018 Mar 5. PMID 29508167
- [Background] Ferrando C, Aguilar G, Piqueras L, Soro M, Moreno J, Belda FJ. Sevoflurane, but not propofol, reduces the lung inflammatory response and improves oxygenation in an acute respiratory distress syndrome model: a randomised laboratory study. Eur J Anaesthesiol. 2013 Aug;30(8):455-63. doi: 10.1097/EJA.0b013e32835f0aa5. PMID 23545542